CLINICAL TRIAL: NCT05237323
Title: The Efficacy and Safety of Mycophenolate Mofetil in the Treatment of Lymphocytic Myocarditis in Comparison With Azathioprine
Brief Title: Micophenolate Mofetil Versus Azathioprine in Myocarditis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122
Record Dates: First submitted 2022-01-13; First posted 2022-02-14 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Lymphocytic Myocarditis (Disorder); Heart Failure; Dilated Cardiomyopathy; Cardiomyopathies; Sudden Cardiac Death
Keywords: virus-negative lymphocytic myocarditis; myocarditis; immunosuppressive therapy; azathioprine; glucocorticosteroids; endomyocardial biopsy; Parvovirus B19; Anticardial antibodies
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated; Cardiomyopathies; Death, Sudden, Cardiac; Myocarditis | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- main group (Experimental): Group 1 included 25 patients who received mycophenolate mofetil 2 g per day per os and methylprednisolone in an average starting dose 24 [24; 32] mg per day per os and standard drug therapy for heart failure (beta-blockers, angiotensin converting enzyme inhibitors or angiotensin II receptor blocker, mineralocorticoid receptor antagonist angiotensin receptor-neprilysin inhibitor (if required), diuretics (if required)).
  Interventions: Drug: mycophenolate mofetil 2 g per day
- control group (Active Comparator): Group 2 included 25 patients who received azathioprine at an average dose of 150 [75; 150] mg per day per os and methylprednisolone in an average starting dose 24 [24; 32] mg per day per os and standard drug therapy for heart failure (beta-blockers, angiotensin converting enzyme inhibitors or angiotensin II receptor blocker, mineralocorticoid receptor antagonist angiotensin receptor-neprilysin inhibitor (if required), diuretics (if required))
  Interventions: Drug: azathioprine of 150 [75; 150] mg per day

INTERVENTIONS:
Drug: mycophenolate mofetil 2 g per day — mycophenolate mofetil 2 g per day and methylprednisolone in an average starting dose 24 [24; 32] mg per day and standard drug therapy for heart failure.
  Arms: main group
Drug: azathioprine of 150 [75; 150] mg per day — azathioprine at an average dose of 150 [75; 150] mg per day and methylprednisolone in an average starting dose 24 [24; 32] mg per day and standard drug therapy for heart failure.
  Arms: control group

SUMMARY:
The study is aimed at studying the direct efficacy of mycophenolate mofetil (mycophenolate mofetil, CellCept, Genentech, N015393/02, 12.08.2009) (in combination with corticosteroids (methylprednisolone, Metypred, Orion, 003467, 26.02.2016)) in the treatment of lymphocytic myocarditis: the effect on symptoms, structural and functional parameters of the heart, on the outcomes of lymphocytic myocarditis: mortality, the need for transplantation, other surgical interventions, the incidence of unwanted side effects, and forced cancellation (replacement) of the drug. To compare the data on the efficacy and safety of therapy with mycophenolate mofetil (in combination with corticosteroids) with the standard regimen of therapy for lymphocytic myocarditis (corticosteroids in combination with azathioprine), including in cases of forced replacement of drugs with each other.

DETAILED DESCRIPTION:
From October 2020 to December 2022, it is planned to enroll 50 patients in "case-control" study diagnosed with virus negative lymphocytic myocarditis at the University Clinical Hospital No. 1, who meet the inclusion criteria. In this study, counting the sample is impossible and such a number of patients is explained by both the rarity of the pathology and the expensive diagnostic endomyocardial biopsy for mandatory confirmation of the diagnosis. Further, the patients will be divided into 2 groups. The main group is methylprednisolone at a starting dose of 24-40 mg / day + mycophenolate 2 g / day per os for 1 month, followed by a decrease in the dose of methylprednisolone to a maintenance dose (4-8 mg / day). The comparison group is methylprednisolone at a starting dose of 24-40 mg / day per os in combination with azathioprine 2 mg / kg per os (100-150 mg / day). All patients will receive standard heart failure therapy including beta-blockers, angiotensin converting enzyme inhibitors or angiotensin II receptor blocker, mineralocorticoid receptor antagonist, angiotensin receptor-neprilysin inhibitor (if required), diuretics (if required).

The first stage is the patient screening (medical history, newly admitted with suspected myocarditis) which includes examination to verify the diagnosis of severe and moderate subacute/chronic myocarditis. Basic research methods: anamnesis, physical examination, blood tests (general, biochemical), electrocardiogram, daily monitoring of electrocardiogram by Holter, transthoracic echocardiography, determination of the level of anticardial antibodies in the blood: regardless of the meal, venous blood is collected in a sterile test tube, then on the same day it is transported under normal conditions to the laboratory of the city clinical hospital №52 for immunomorphological examination. Reference values: antibodies to antigens of cardiomyocyte nuclei (no antibody titer), antibodies to endothelial antigens (antibody titer 1:40), antibodies to cardiomyocyte antigens (antibody titer 1:40), antibodies to smooth muscle antigens (antibody titer 1:40), antibodies to the antigens of the fibers of the cardiac conduction system (antibody titer 1:40) Endomyocardial biopsy of the right ventricle with determination of the genome of cardiotropic viruses in the myocardium by polymerase chain reaction, standard histological examination (staining with hematoxylin-eosin, according to Van Gieson), immunohistochemistry-specific antibodies for leukocytes (CD45), macrophages (CD68), T cells (CD3) and their main subtypes, helper (CD4) and cytotoxic (CD8) cells, and B cells (CD19/CD20): quantitative criteria to improve the diagnostic yield of endomyocardial biopsy in myocarditis include the Marburg criteria, based on the presence of >14 mononuclear leukocytes/mm2 on bioptic samples, with the presence of >7 T lymphocytes per mm2. These criteria were adopted in a position statement by the European Society of Cardiology experts). Additionally (for special indications): multislice computer tomography scanning and / or magnetic resonance imaging of the heart with intravenous contrasting with gadolinium (CAS: 88344-16-5), coronary angiography and myocardial scintigraphy (for patients with suspected coronary artery disease, high pretest likelihood of coronary heart disease more than 65%, positive exercise test, coronary atherosclerosis on computed tomography or previous myocardial infarction), genetic counseling (the process of genetic counseling is about sharing information regarding genetic and disease risks in a manner useful to an individual, couple, or family copes with a possible cause of genetically determined heart diseases: hypertrophic cardiomyopathy, arrhythmogenic right ventricular dysplasia, canalopathy or restrictive cardiomyopathy).

Endomyocardial biopsy is performed according to indications developed in the clinic and consistent with the European recommendations for myocardial biopsy (2007).

At the second stage, patients who confirmed virus-negative lymphocytic myocarditis during endomyocardial biopsy, are included in the study according to the inclusion and non-inclusion criteria. All patients sign informed consent to participate in the study. The second stage involves the determination of indications for the appointment of immunosuppressive therapy (verified diagnosis of severe and moderate myocarditis, resistance to standard cardiotropic therapy for 2 months, the absence of markers of active viral infection in the blood and viral genome in the myocardium (adenovirus, enterovirus, citomegalovirus, Epstein-Barr virus, human herpes virus 6, hepatitis C virus, the human immunodeficiency virus, influenza, coronavirus (MERS-CoV, SARS-CoV, SARS-CoV-2), with the exception of parvovirus B19, the absence of other active infection). The distribution into two groups is made by the researcher. All patients are matched by gender and age. If the patient has previously received azathioprine with insufficient effect or side effects were present, then the patient is included in the main group and vice versa. The observation period is at least 6 months. The frequency of control examinations: 2 months after the start of therapy (with a stable course of myocarditis, studies are performed in absentia): blood tests (general, biochemical), electrocardiogram, 24 hour monitoring of electrocardiogram by Holter, transthoracic echocardiography, determination of the level of anticardial antibodies in the blood) and then every 6 months (with a stable course of myocarditis, studies are performed in absentia): blood tests (general, biochemical), electrocardiogram, daily monitoring of electrocardiogram by Holter, transthoracic echocardiogram, determination of the level of anticardial antibodies in the blood). observation median - one year. Statistical processing: SPSS version 23 software package.

Qualitative, quantitative variables:

Discrete data will be presented in the form of absolute values and percentages, continuous data - in the form of arithmetic mean ± standard deviation in the case of normal distribution or in the form of quartiles 50 [25; 75], if the distribution differs from normal.

Determination of the type of distribution:

To assess the normality of the distribution, the Kolmogorov-Smirnov test will be used.

Comparison of indicators between groups depending on the type of distribution:

Comparison of patients by groups will be carried out using χ2 or Fisher's exact test for categorical dichotomous variables, for the rest - using the Student's t-test (with a normal distribution and the number of observations over 25) or Mann-Whitney U-test.

Survival assessment:

Survival analysis will be performed with Kaplan-Meier curves.

Regression analysis:

Correlation analysis followed by linear regression will be performed to identify possible predictors of outcomes.

Differences will be considered significant at a significance level of p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Presence of written informed consent of the patient to participate in the study;
* Age 18 and older;
* The diagnosis of myocarditis, established using endomyocardial biopsy (active or borderline myocarditis according to Dallas criteria, virus negative, excluding parvovirus B19);
* Chronic heart failure 2-4 according to New York Heart Association functional classification;
* Signs of left ventricular dysfunction, persisting after 2 months of optimal drug therapy (therapy for heart failure, including angiotensin-converting enzyme inhibitors or angiotensin II receptor blockers, beta-blockers, mineralocorticoid receptor antagonists, diuretics, angiotensin receptors and neprilysin inhibitors): end-diastolic the size of the left ventricle is more than 5.5 cm, the ejection fraction is less than 50%;

Non-inclusion criteria:

* History of myocardial infarction/acute coronary syndrome.
* Chronic ischemic heart disease with hemodynamically significant stenoses of the coronary arteries (70% or more).
* Congenital heart defects.
* History of infective endocarditis less than 6 months old.
* Thyrotoxic heart.
* Hypertensive heart (left ventricular hypertrophy more than 14 mm).
* Hypertrophic cardiomyopathy.
* Verified amyloidosis, sarcoidosis, other storage diseases.
* Diffuse connective tissue diseases.
* Verified systemic vasculitis.
* Lymphoproliferative diseases.
* Condition after chemotherapy with anthracycline drugs.
* Heart surgery less than 2 months old.

Exclusion Criteria:

* Patient refusal to participate in the study;
* Pregnancy;
* Inability to adequately control therapy and follow the research protocol (serious mental disorders, remoteness of residence, non-compliance of the patient)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
cardiovascular death | From the start of therapy for at least one year or until the patient's death
  frequency of biological death from cardiovascular causes of a patient recorded in a hospital or at home, confirmed by a death certificate (with or without autopsy results); the relevant information was obtained directly from the relatives of the deceased.
heart transplant | From the start of therapy for at least one year or until the patient's death
  frequency of heart transplantation due to lack of effect from immunosuppressive therapy and standard cardiotropic therapy with persistent heart failure of NYHA functional class 4 requiring constant inotropic or circulatory support or Intractable life-threatening arrhythmias unresponsive to medical therapy, catheter ablation, surgery, and/or implantable cardioverter-defibrillator.

SECONDARY OUTCOMES:
Dynamics of heart failure in accordance with New York Heart Association classification | up to 1 week, 2 months after therapy, then 6 months later
  assessment of the dynamics of the severity of the condition according to the classification of the functional classification of the New York Heart Association using the test with a six-minute walk
dynamics of left ventricle ejection fraction | up to 1 week
  dynamics of left ventricle ejection fraction by Simpson technique according to transthoracic echocardiography
dynamics of left ventricle ejection fraction | 2 months after starting therapy
  dynamics of left ventricle ejection fraction by Simpson technique according to transthoracic echocardiography
dynamics of left ventricle ejection fraction | 6 months after starting therapy
  dynamics of left ventricle ejection fraction by Simpson technique according to transthoracic echocardiography
dynamics of the end-diastolic diameter of the left ventricle (cm) | up to 1 week
  dynamics of left end-diastolic diameter of the left ventricle (cm) according to transthoracic echocardiography
dynamics of the end-diastolic diameter of the left ventricle (cm) | 2 months after starting therapy
  dynamics of left end-diastolic diameter of the left ventricle (cm) according to transthoracic echocardiography
dynamics of the end-diastolic diameter of the left ventricle (cm) | 6 months after starting therapy
  dynamics of left end-diastolic diameter of the left ventricle (cm) according to transthoracic echocardiography
dynamics of the end-diastolic volume of the left ventricle (ml) | up to 1 week
  dynamics of the end-diastolic volume of the left ventricle (ml) according to transthoracic echocardiography
dynamics of the end-diastolic volume of the left ventricle (ml) | 2 months after starting therapy
  dynamics of the end-diastolic volume of the left ventricle (ml) according to transthoracic echocardiography
dynamics of the end-diastolic volume of the left ventricle (ml) | 6 months after starting therapy
  dynamics of the end-diastolic volume of the left ventricle (ml) according to transthoracic echocardiography
dynamics of the end-systolic volume of the left ventricle (ml) | up to 1 week
  dynamics of the end-systolic volume of the left ventricle (ml) according to transthoracic echocardiography
dynamics of the end-systolic volume of the left ventricle (ml) | 2 months after starting therapy
  dynamics of the end-systolic volume of the left ventricle (ml) according to transthoracic echocardiography
dynamics of the end-systolic volume of the left ventricle (ml) | 6 months after starting therapy
  dynamics of the end-systolic volume of the left ventricle (ml) according to transthoracic echocardiography
dynamics of the systolic pressure in the pulmonary artery according to transthoracic echocardiography data. | up to 1 week
  Change in systolic pressure in the pulmonary artery (mm Hg) in comparison with baseline values (at the time of inclusion in the study
dynamics of the systolic pressure in the pulmonary artery according to transthoracic echocardiography data. | 2 months after starting therapy
  Change in systolic pressure in the pulmonary artery (mm Hg) in comparison with baseline values (at the time of inclusion in the study
dynamics of the systolic pressure in the pulmonary artery according to transthoracic echocardiography data. | 6 months after starting therapy
  Change in systolic pressure in the pulmonary artery (mm Hg) in comparison with baseline values (at the time of inclusion in the study
drug withdrawal | up to 1 week
  frequency of drug withdrawal due to side effects: myelodepression (leukopenia, thrombocytopenia, anemia), development of secondary infections, megaloblastic erythropoiesis and macrocytosis, nausea, vomiting, anorexia, skin rash, arthralgia, myalgia, erosive and ulcerative lesions of the oral cavity, medicinal, cholestatic hepatitis, toxic hepatitis or no effect according to transthoracic echocardiography (left ventricle ejection fraction, size of the left ventricle, systolic pressure in the pulmonary artery) and anticardial antibodies.
drug withdrawal | 2 months after starting therapy
  frequency of drug withdrawal due to side effects: myelodepression (leukopenia, thrombocytopenia, anemia), development of secondary infections, megaloblastic erythropoiesis and macrocytosis, nausea, vomiting, anorexia, skin rash, arthralgia, myalgia, erosive and ulcerative lesions of the oral cavity, medicinal, cholestatic hepatitis, toxic hepatitis or no effect according to transthoracic echocardiography (left ventricle ejection fraction, size of the left ventricle, systolic pressure in the pulmonary artery) and anticardial antibodies.
drug withdrawal | 6 months after starting therapy
  frequency of drug withdrawal due to side effects: myelodepression (leukopenia, thrombocytopenia, anemia), development of secondary infections, megaloblastic erythropoiesis and macrocytosis, nausea, vomiting, anorexia, skin rash, arthralgia, myalgia, erosive and ulcerative lesions of the oral cavity, medicinal, cholestatic hepatitis, toxic hepatitis or no effect according to transthoracic echocardiography (left ventricle ejection fraction, size of the left ventricle, systolic pressure in the pulmonary artery) and anticardial antibodies.
drug replacement due to side effect | up to 1 week
  frequency of drug replacement due to side effect: myelodepression (leukopenia, thrombocytopenia, anemia), development of secondary infections, megaloblastic erythropoiesis and macrocytosis, nausea, vomiting, anorexia, skin rash, arthralgia, myalgia, erosive and ulcerative lesions of the oral cavity, medicinal , cholestatic hepatitis, toxic hepatitis or no effect according to ECHO-KG (Ejection fraction, size of the left ventricle, systolic pressure in the pulmonary artery) and anticardial antibodies
drug replacement due to side effect | 2 months after starting therapy
  frequency of drug replacement due to side effect: myelodepression (leukopenia, thrombocytopenia, anemia), development of secondary infections, megaloblastic erythropoiesis and macrocytosis, nausea, vomiting, anorexia, skin rash, arthralgia, myalgia, erosive and ulcerative lesions of the oral cavity, medicinal , cholestatic hepatitis, toxic hepatitis or no effect according to ECHO-KG (Ejection fraction, size of the left ventricle, systolic pressure in the pulmonary artery) and anticardial antibodies
drug replacement due to side effect | 6 months after starting therapy
  frequency of drug replacement due to side effect: myelodepression (leukopenia, thrombocytopenia, anemia), development of secondary infections, megaloblastic erythropoiesis and macrocytosis, nausea, vomiting, anorexia, skin rash, arthralgia, myalgia, erosive and ulcerative lesions of the oral cavity, medicinal , cholestatic hepatitis, toxic hepatitis or no effect according to ECHO-KG (Ejection fraction, size of the left ventricle, systolic pressure in the pulmonary artery) and anticardial antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan S Rud', Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Bol'shaya Pirogovskaya Street 6, 1 Building ,, Russia

IPD SHARING:
Plan to Share IPD: No
The provision of data is possible only upon official request.

REFERENCES:
- See also: Related Info — https://russjcardiol.elpub.ru/jour/article/view/4650